CLINICAL TRIAL: NCT04859881
Title: Risk Factors Associated With Barotrauma in COVID-19 Patients
Brief Title: Risk Factors for Barotrauma in COVID-19
Status: Completed | Type: Observational
Sponsor: Hospital General Ajusco Medio (Other)
Collaborators: Horacio Marquez-Gonzalez (Unknown); Carlos Torruco-Sotelo (Unknown); Sebastian Rodriguez-Llamazares (Unknown)
Responsible Party: Principal Investigator, Karla Verónica Chavez-Tostado, Head of Surgery Department, Hospital General Ajusco Medio
Other Study IDs: HGAM01
Record Dates: First submitted 2021-04-19; First posted 2021-04-26 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Barotrauma; Covid19
Keywords: Barotrauma; COVID-19
MeSH Terms: conditions — Barotrauma; COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Barotrauma/cases: Cases were defined as patients with barotrauma consulted with the Surgery Department
  Interventions: Other: No intervention
- No braotruma/Controls: Controls were selected from a random sample of the COVID-19-ARDS cohort.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Barotrauma in mechanical ventilation (MV) is defined as lung damage attributable to the application of high airway pressure and is one of the potential mechanisms of ventilator-induced lung injury (VILI). Previous studies have shown an increased mortality in patients with barotrauma under MV; pneumothorax (PTX) being the most common presentation, but it can also present as pneumomediastinum (PM) with or without PTX, with extension to soft tissue as subcutaneous emphysema or even as pneumo-retroperitoneum and pneumo-scrotum.

Traditionally, underlying lung disease or age are known risk factors for non-trauma related barotrauma. However, in patients with novel coronavirus disease (COVID-19), the incidence of this complication is more common than in non-infected patients, as recently reported. Since little is known regarding which are the main risk factors for these events to develop, most pathophysiological mechanisms remain unexplained.

The aim of this study was to determine the risk factors for developing barotrauma in patients under MV with COVID-19 associated Acute Respiratory Distress Syndrome (ARDS). Secondary objectives were to determine the incidence of barotrauma and its association with mortality.

ELIGIBILITY:
Inclusion Criteria:

* Patients under MV fulfilling the Berlin definition for ARDS, with positive SARS-COV2 real time polymerase chain reaction

Exclusion Criteria:

* Incomplete clinical records and other causes of extrapulmonary air

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diagnosis of severe SARS-COV2 infection and mechanical ventilation, admitted in a single-center community Hospital in Mexico City.
Sampling Method: Non-Probability Sample
Enrollment: 262 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Barotrauma development | During patient hospitalization, an average of one month
  Diagnosis of barotrauma in patients under mechanical ventilation with COVID-19 associated Acute Respiratory Distress Syndrome

SECONDARY OUTCOMES:
Mortality | During patient hospitalization, an average of one month
  Dead of patient

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital General Ajusco Medio, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No